CLINICAL TRIAL: NCT01376999
Title: Step Up Versus Step Down in Controlled Ovarian Stimulation for Intrauterine Insemination. A Controlled Randomised Trial.
Brief Title: Step Up Versus Step Down in Controlled Ovarian Stimulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Miguel Angel Checa, MD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UREP-01-2009
Record Dates: First submitted 2011-06-17; First posted 2011-06-20 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: No Explained Sterility
Keywords: Sterility; FSH-r; intrauterine insemination; unexplained sterility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Step Down (Experimental): Step Down: We begin the COS (controlled ovarian stimulation) with 150 IU of FSH-r until 7th day of stimulation. This day we make an adjustment reducing the dose if necessary.
  Interventions: Drug: FSH-r (Follicule stimulate hormone)
- Step Up (Active Comparator): Step up: We begin the COS (controlled ovarian stimulation) with 75 IU of FSH-r until 7th day of stimulation.This day we make an adjustment increasing the dose if necessary.
  Interventions: Drug: FSH-r (Follicule stimulate hormone)

INTERVENTIONS:
Drug: FSH-r (Follicule stimulate hormone) — Step-Up: 75 IU FSH-r Step-Down: 150 FSH-r

SUMMARY:
The aim of the study is to evaluate if the Step up protocol is equal or superior regarding efficacy and security than the step down protocol. In couple submitted two intrauterine insemination.

ELIGIBILITY:
Inclusion Criteria:

* Women with unexplained sterility with needs of intrauterine insemination.

Exclusion Criteria:

* Contraindications to intrauterine insemination.

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 158 (Actual)
Dates: Start 2010-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Ovulation rate | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Spain

REFERENCES:
- [Derived] Robles A, Gayete-Lafuente S, Prat M, Gonzalez-Comadran M, Checa MA. The step-up protocol increases clinical pregnancy rates compared with the step-down in patients with unexplained infertility. A randomized controlled trial. JBRA Assist Reprod. 2022 Nov 9;26(4):599-605. doi: 10.5935/1518-0557.20210112. PMID 35243855